CLINICAL TRIAL: NCT06824337
Title: Effect of Targeted Mobilization Program Applied After Caesarean Section Surgery on Care Outcomes: Randomized Controlled Study
Brief Title: Effect of Targeted Mobilization Program
Acronym: Mobilization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22504254-050.04
Record Dates: First submitted 2024-12-18; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-12

CONDITIONS: Caesarean Section; Mobility; Pain; Breastfeeding
Keywords: Caesarean section; mobilization; pain; breastfeeding
MeSH Terms: conditions — Pain; Breast Feeding

STUDY DESIGN:
Intervention Model Description: The research is a two-group parallel randomized controlled experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The first interview with the intervention group patients will be held when the patients arrive at the hospital. In these interviews, the patients will first be introduced to the patients, detailed information will be provided about the research, their verbal/written informed consent will be obtained, and answers will be obtained to the questions in the patient information form. In addition, the content of the early mobilization training given to the patients in the first interview, what early mobilization is, why it is important, what benefits it provides, what the mobilization goals determined for the patient within the scope of the research are, the benefits of walking and the expected results will be explained. It will be explained how to benefit from the smartphone during the mobilization process. In addition to all the training, the patients in the intervention group will be given detailed information about what they need to record in the mobilization diary (total time they walke
  Interventions: Other: mobilization training and targeted mobilization
- control group (No Intervention): Women in the control group will be left to the routine care of the institution. Within the scope of routine care, women in this group will be asked to record their walking distance.

INTERVENTIONS:
Other: mobilization training and targeted mobilization — In the first interview with the patients, the content of the early mobilization training given to the patients, what early mobilization is, why it is important, what benefits it provides, what the mobilization goals determined for the patient within the scope of the research, the benefits of walking and the expected results will be explained. It will be explained how to benefit from the smartphone during the mobilization process. In addition to all the training, the patients in the intervention group will be given detailed information about what they need to record in the mobilization diary (total time they walked, how many steps they took in the pedometer application after each mobilization, positive/negative situations they experienced while standing up and walking) and all the forms that will be used in the data collection phase.
  Arms: Experimental group

SUMMARY:
This study was planned to evaluate the effect of early mobilization training given to patients undergoing cesarean section in the preoperative period and targeted mobilization program applied after the surgery, on preventing gastrointestinal complications that may develop after the surgical intervention and participating in breastfeeding and baby care. The research will be conducted in experimental design. The research will begin after receiving written permission from Niğde Ömer Halisdemir University Ethics Committee, Niğde Provincial Health Directorate and Ömer Halisdemir Training and Research Hospital. Pregnant women who are between the ages of 18-35, who are at least a primary school graduate, who gave birth at term, who have a live singleton pregnancy, and who do not have a risky pregnancy history (DVT, thromboembolism) will be included in the study. Before starting the research, the study will begin by obtaining institutional permissions and written permission from the pregnant women. Personal Information Form prepared in line with the literature, postoperative gastrointestinal functions information form, postoperative abdominal distension diagnosis form, walking chart, VAS, LATCH Breastfeeding Diagnosis and Evaluation Scale and Breastfeeding Information Form data collection forms will be used to collect data. The data will be evaluated on a computer using the IBM SPSS Statistics 24 (Statistical Package for the Social Sciences for Windows) package program. Appropriate statistical analyzes will be used to evaluate the data

DETAILED DESCRIPTION:
Cesarean section is life-saving for the mother and baby when necessary, but it can increase maternal mortality and morbidity rates when compared to vaginal birth. Cesarean section rates are increasing by 4% each year in the world. FIGO which took place in Brazil in 2018, reported that cesarean section rates doubled between 2000 and 2015, revealing a serious problem globally . When cesarean section rates were compared between 2000 and 2015, it was determined that they increased from 19.6% to 26.9% in Western Europe, from 32.3% to 44.3% in Latin America, and from 7.2% to 18.1% in South Asia. The cesarean section rate in Turkey was 21.2% in 2003, 36.7% in 2008, and increased to 48.5% in 2013. The significant increase in the number of cesarean sections performed each year worldwide has made postoperative care even more important. As in all abdominal surgeries, delayed gas release, delayed return of bowel movements, delayed resumption of oral intake, wound healing, urinary retention, atalactasia, bleeding, adhesion, hematoma, thrombophlebitis, venous and pulmonary embolism, coagulopathies, and anesthesia-related problems are observed after cesarean surgery. In addition, problems such as failure to participate in baby care and delay in starting breastfeeding are also encountered. Early mobilization is very valuable to prevent these complications, and studies argue that early mobilization can prevent negative outcomes related to many systems in the body. In the ERAS guideline created specifically for patients undergoing cesarean section, although it is stated that there are no randomized controlled trials with strong methodology regarding early mobilization, it is recommended that patients after cesarean section should also be mobilized early (Very low-level evidence, weak recommendation). Although early mobilization is considered an important element of postoperative care, it is not yet fully known how to best implement it in clinical practice. Because there are limited scientific studies in the literature supporting the superiority of any mobilization program over another. The independent positive contributions of early mobilization to postoperative patient outcomes are accepted, the importance of timing is emphasized, but there is not yet sufficient evidence regarding the effect of frequency and duration on patient outcomes, there is a need for scientific studies emphasizing the importance of an early mobilization plan structured with daily written goals starting from the day of surgery, including getting out of bed and walking distances. In preoperative patient education, determining postoperative step goals and using a pedometer to achieve these goals and/or keeping a mobilization diary are stated as other practices that can increase patients' compliance with postoperative mobilization programs. The participation of nurses, who are involved in all processes of surgery, in the patient education phase is also very important and nurses should be the most competent team members in the implementation of standardized early mobilization protocols. Therefore, nurses should focus on developing and implementing protocols that aim to minimize the dependency of hospitalized patients on nurses, encourage mobilization, and prevent a decrease in functionality. Thus, nurses will be able to assume more roles and responsibilities in ensuring early mobilization. No study has been found in the literature in which a targeted mobilization program was implemented in cesarean surgery. In this context, the study is planned to evaluate the effect of early mobilization education given to patients undergoing cesarean section in the preoperative period and the targeted mobilization program applied after surgery on preventing gastrointestinal complications that may develop after surgery and participating in breastfeeding and baby care.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,
* At least primary school graduate,
* Giving birth at term
* Having a live singleton pregnancy,
* No risky pregnancy history (DVT, thromboembolism)
* Women who can use a mobile phone

Exclusion Criteria:

* Exclusion Criteria for the Study
* Those who want to leave the study,
* Undergoing emergency caesarean section,
* Not recording walking distance
* Women who cannot be interviewed within 24 hours of discharge
* Women who develop maternal or neonatal complications after birth

Ages: 18 Months to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — primipara women
Enrollment: 64 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Gastrointestinal Functions Information Form | 3 month
  The form, which will evaluate women's postoperative GI functions, includes six questions that evaluate the time and amount of oral intake after surgery, the time of first gas and defecation, and nausea and vomiting.
Postoperative Abdominal Distension Diagnosis Form | 3 month
  The form is a measurement tool that evaluates abdominal distension status at 6, 12, 24 and 48 hours after surgery using a scale ranging from 0 (no distension) to 10 (the most severe distension possible)
VAS (Visual Analog Scala) | 3 month
  It consists of a 10 cm long horizontal or vertical line, which is often used to measure subjective parameters. One end of the line indicates 0 = "no pain", the other 10 = worst/unbearable pain.

SECONDARY OUTCOMES:
LATCH Breastfeeding Diagnostic and Assessment Scale | 3 month
  Each criterion that makes up the LATCH Breastfeeding Diagnosis and Assessment Scale is given a score of 0, 1, or 2. Breastfeeding success is assessed by adding the scores. The highest score that can be obtained from the scale is 10 and the lowest score is 0.
Breastfeeding Information Form | 3 month
  The form consists of six questions to determine the breastfeeding status, frequency and participation in baby care of women on days 0, 1 and 2 after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: isa temur, Dr, Principal Investigator — NİĞDE ÖMER HALİSDEMİR UNIVERCITY
Locations (1):
- Niğde Ömer Halisdemir Univercity, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No